CLINICAL TRIAL: NCT01816243
Title: Evaluation Study of Efficacy and Safety of TTS-Fentanyl in Chronic Non-Malignant Pain
Brief Title: An Efficacy and Safety Study of Transdermal Therapeutic System (TTS)-Fentanyl in Thai Participants With Chronic Non-Malignant Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR009925; DURO-THAI-3
Record Dates: First submitted 2013-03-19; First posted 2013-03-22 (Estimated); Results first posted 2013-06-11 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Chronic Non-Malignant Pain; TTS-fentanyl; Durogesic
MeSH Terms: conditions — Chronic Pain | interventions — Fentanyl; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transdermal Therapeutic System (TTS)-fentanyl (Experimental): Transdermal Therapeutic System (TTS)-fentanyl patches releasing fentanyl in the range of 12.5 to 100 microgram per hour (mcg/hr) rate. The initial dose of fentanyl TTS will be calculated based on each participant's opioid requirement. Patches will be usually replaced every 72 hours. Doses will be escalated in steps of 25 mcg/hr, if pain cannot be controlled. Oral morphine syrup is allowed to titrate the dose of TTS-fentanyl. The study duration will be 30 days after first patch application.
  Interventions: Drug: TTS-Fentanyl; Drug: Morphine

INTERVENTIONS:
Drug: TTS-Fentanyl — Transdermal Therapeutic System (TTS)-fentanyl patches releasing fentanyl in the range of 12.5 to 100 microgram per hour (mcg/hr) rate. The initial dose of fentanyl TTS will be calculated based on each participant's opioid requirement. Patches will be usually replaced every 72 hours. Doses will be escalated in steps of 25 mcg/hr, if pain cannot be controlled. The study duration will be 30 days after first patch application.
  Other Names: Durogesic
Drug: Morphine — Participants will be allowed the use of oral morphine syrup for the duration of TTS-fentanyl treatment to enable appropriate dose titration. It is expected that most of the participants will be titrated to an appropriate dose of TTS-fentanyl within 1 week.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Transdermal Therapeutic System (TTS)-fentanyl patch (transdermal patch containing a drug that is put on the skin so the drug will enter the body through the skin) in Thai participants with chronic (lasting a long time) non-malignant (non-cancerous) pain.

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention), single arm study to assess the efficacy and safety of TTS-fentanyl in Thai participants with chronic non-malignant pain (except for headaches or central spinal cord mediated pain). The study will consist of 2 phases: stabilization phase (up to 7 days before starting the treatment) and treatment phase (30 days). The first patch will be applied by Investigator then by participants themselves until 30 days. All participants will start the treatment with patch releasing 25 micrograms per hour (mcg/h) of fentanyl . The patches will be replaced every 3 days. On Day 3, and every 3 days thereafter, the TTS-fentanyl dose can be titrated (slow increase in drug dosage, guided by participant's responses) as per participant's need. The duration of the treatment will be 30 days after first patch application. The dose of TTS-fentanyl can be slowly increased if needed, by 25 mcg/h to achieve adequate pain control. No increase in TTS-fentanyl dose will be performed within the 72-hour dosing interval. Participants will be allowed the use of oral morphine syrup for the duration of TTS-fentanyl treatment to enable appropriate TTS-fentanyl dose titration. Primary efficacy assessment will be pain control rated by participants. Assessment time points will be Day 0 (Baseline), Day 15 and Day 30 (trial end). At the end of study, global preference on efficacy, side effects and overall satisfaction will also be rated by Investigator and participants. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic non-malignant pain (of any etiology except for headaches or central spinal cord mediated pain) with moderate (medium level of seriousness) to severe (very serious, life threatening) pain that requires treatment with a potent opioid
* Participants must also be currently treated with short or long acting opioid medications other than Transdermal Therapeutic System (TTS)-fentanyl at a dose less than or equal to 134 milligram per day (mg/day) of oral morphine (or an equianalgesic dose of another opioid), participants may have been treated with TTS-fentanyl in the past
* Participants who had side effects after receiving Non Steroidal Anti-inflammatory Drugs (NSAIDs)
* Participants who failed from other treatments such as operation or lack of efficacy of current treatment
* Participants with spinal cord stimulators may enroll, provided that they turn the spinal cord stimulator off for the duration of the trial, or leave it continually on for the duration of the trial

Exclusion Criteria:

* History of allergy, hypersensitivity, or lack of ability to tolerate fentanyl
* Skin disease that precludes the use of the transdermal system or which could affect the absorption of fentanyl or local tolerability
* History or suspicion of alcohol or drug abuse within the past 5 years
* History of narcotic (strong habit-forming drug that stops pain and depresses the central nervous system) therapy
* Pregnancy or breast-feeding female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd.,Thailand Clinical Trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (2):
- Thailand (2):
  - Department of Anesthesia, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok
  - Bangkok

RESULTS

PARTICIPANT FLOW:
Groups:
- Transdermal Therapeutic System (TTS) - Fentanyl: Transdermal Therapeutic System (TTS) - fentanyl patches releasing fentanyl in the range of 12.5 to 100 microgram per hour (mcg/hr) rate. The initial dose of fentanyl TTS was calculated based on each participant's opioid requirement. Patches were usually replaced every 72 hours. Doses were escalated in steps of 25 mcg/hr, if pain cannot be controlled. 90 milligram per day (mg/day) of oral morphine was allowed as supplementary analgesic. The study duration was 30 days after first patch application.
Period: Overall Study
Arm/Group | Transdermal Therapeutic System (TTS) - Fentanyl
Started | 39
Completed | 27
Not Completed | 12
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1
Not completed — Not eligible for the study | 1
Not completed — Amputation | 3

BASELINE CHARACTERISTICS:
Population: The demographics was reported for only 38 participants who were eligible for the study.
Arm/Group | Transdermal Therapeutic System (TTS) - Fentanyl
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.39 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 23
Pain Intensity Rating [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was assessed on 11-point Numeric Rating Scale (NRS); score ranges from 0 to 10, where 0=no pain and 10=worst pain.
  units on a scale | 6.54 (2.02)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Intensity Rating at Day 15
Description: Pain intensity was assessed on 11-point Numeric Rating Scale (NRS); score ranges from 0 to 10 where 0=no pain and 10=worst pain.
Time Frame: Baseline and Day 15
Population: Intent-to-treat (ITT) population set included all participants who received at least one dose of study medication and who had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Transdermal Therapeutic System (TTS) - Fentanyl
Number analyzed (Participants) | 37
Units on a scale | -1.56 (3.15)

2. Primary Outcome: Change From Baseline in Pain Intensity Rating at Day 30
Description: Pain intensity was assessed on 11-point NRS; score ranges from 0 to 10 where 0=no pain and 10=worst pain.
Time Frame: Baseline and Day 30
Population: The ITT population set included all participants who received at least one dose of study medication and who had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Transdermal Therapeutic System (TTS) - Fentanyl
Number analyzed (Participants) | 37
Units on a scale | -1.95 (3.28)

3. Secondary Outcome: Number of Participants With Investigator's Global Assessment
Description: Investigator would complete a global assessment of the participants treatment with respect to pain control using a 9-point scale (-4 to 4; where, -4=100 percent (%) worse, 0=unchanged and 4=100% improvement), safety using 5-point scale (1 to 5; where, 1=no, 2=mild, 3=moderate, 4=severe and 5=most severe side effects) and 5-point overall satisfaction scale (1-5; where, 1=no, 2=mild, 3=moderate, 4=good, 5=excellent). Number of participants with Investigator's assessment with respect to efficacy, safety and overall satisfaction were reported.
Time Frame: Day 30
Population: The ITT population set included all participants who received at least one dose of study medication and who had at least one post-baseline efficacy assessment. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Participants
Arm/Group | Transdermal Therapeutic System (TTS) - Fentanyl
Number analyzed (Participants) | 27
Participants
  Efficacy, 100% Worse | 0
  Efficacy, 75% Worse | 0
  Efficacy, 50% Worse | 1
  Efficacy, 25% Worse | 0
  Efficacy, Unchanged | 7
  Efficacy, 25% Improve | 2
  Efficacy, 50% Improve | 6
  Efficacy, 75% Improve | 4
  Efficacy, 100% Improve | 7
  Safety, No | 16
  Safety, Mild | 9
  Safety, Moderate | 2
  Safety, Severe | 0
  Safety, Most severe | 0
  Overall Satisfaction, No | 1
  Overall Satisfaction, Mild | 7
  Overall Satisfaction, Moderate | 6
  Overall Satisfaction, Severe | 8
  Overall Satisfaction, Most Severe | 5

4. Secondary Outcome: Number of Participants With Participant's Global Assessment
Description: Participants global assessment with respect to pain control using a 9-point scale (-4 to 4; where, -4=100% worse, 0=unchanged and 4=100% improvement), safety using 5-point scale (1 to 5; where, 1=no, 2=mild, 3=moderate, 4=severe and 5=most severe side effects) and 5-point overall satisfaction scale (1-5; where, 1=no, 2=mild, 3=moderate, 4=good, 5=excellent). Number of participants with participant's global assessment with respect to efficacy, safety and overall satisfaction were reported.
Time Frame: Day 30
Population: The ITT population set included all participants who received at least one dose of study drug and had at least one post-baseline efficacy assessment. 'N' (number of participants analyzed) = participants who were evaluable for this measure and 'n' = participants who were evaluable for this measure at given time points.
Measure: Number; unit: Participants
Arm/Group | Transdermal Therapeutic System (TTS) - Fentanyl
Number analyzed (Participants) | 34
Participants
  Efficacy, 100% Worse (n=34) | 1
  Efficacy, 75% Worse (n=34) | 0
  Efficacy, 50% Worse (n=34) | 2
  Efficacy, 25% Worse (n=34) | 1
  Efficacy, Unchanged (n=34) | 4
  Efficacy, 25% Improve (n=34) | 13
  Efficacy, 50% Improve (n=34) | 11
  Efficacy, 75% Improve (n=34) | 1
  Efficacy, 100% Improve (n=34) | 1
  Safety, No (n=27) | 16
  Safety, Mild (n=27) | 9
  Safety, Moderate (n=27) | 2
  Safety, Severe (n=27) | 0
  Safety, Most severe (n=27) | 0
  Overall Satisfaction, No (n=27) | 1
  Overall Satisfaction, Mild (n=27) | 7
  Overall Satisfaction, Moderate (n=27) | 6
  Overall Satisfaction, Severe (n=27) | 8
  Overall Satisfaction, Most Severe (n=27) | 5

ADVERSE EVENTS:
Time Frame: From first dose of study medication up to Day 30
Arm/Group | Transdermal Therapeutic System (TTS) - Fentanyl
Serious Adverse Events (participants affected / at risk) | 1/39
Other Adverse Events (participants affected / at risk) | 25/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transdermal Therapeutic System (TTS) - Fentanyl (N=39)
Septic shock (Infections and infestations) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transdermal Therapeutic System (TTS) - Fentanyl (N=39)
Flu-like symptom (General disorders) | 1
Palpitation (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 3
Drowsiness (Nervous system disorders) | 6
Dullness (Nervous system disorders) | 1
Insomnia (Nervous system disorders) | 1
Nightmare (Nervous system disorders) | 1
Hypotension (Cardiac disorders) | 1
Peripheral neuropathy (Nervous system disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 5
Angular ulcer (Skin and subcutaneous tissue disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 8
Non pitting edema (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4

LIMITATIONS AND CAVEATS:
Some limitations of this study were non randomization and uncontrolled design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Timing and publication of the results will be subject to mutual agreement in the project between all Investigators participating in the project and Janssen-Cilag., Thailand.

All manuscripts and abstracts utilizing the data from this study are subjected to the approval of Janssen. All manuscripts and abstract must be sent to Janssen at least one month prior to the submission for publication or presentation.